CLINICAL TRIAL: NCT04929158
Title: Comparison of Clinical Outcomes of Intravascular Ultrasound (IVUS) -Guided and Angiography-Guided Primary Percutaneous Intervention (PCI) in Patients With Acute ST Segment Elevated Myocardial Infarction (STEMI)
Brief Title: Comparison of Clinical Outcomes of IVUS -Guided and Angiography-guided PCI in Patients With Acute STEMI
Status: Available | Type: Expanded Access
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Zhejiang University (Other); First Affiliated Hospital of Wenzhou Medical University (Other); Taizhou First People's Hospital (Other); Changxing People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: clinical 2020-401
Record Dates: First submitted 2021-06-07; First posted 2021-06-18 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: ST Elevation Myocardial Infarction
Keywords: ST Elevation Myocardial Infarction，
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Procedure: Intravascular Ultrasound (IVUS) -guided Primary Percutaneous Intervention (PCI) — Preoperative criminal vascular assessment； The criminal vascular assessment after surgery
  Other Names: Angiography-guided Primary Percutaneous Intervention (PCI)

SUMMARY:
To compare the long-term clinical outcomes of IVUS-guided vs angiography-guided PCI in patients with acute STEMI

DETAILED DESCRIPTION:
This study is a prospective, multicenter, randomized controlled trial, led by the second hospital affiliated to zhejiang university school of medicine, A total of 10 hospitals in zhejiang province interventional cardiovascular center to participate in, plan to recruit 200 STEMI patients.

Subjects according to the proportion of 1:1 were randomly allocated to two treatment groups.(Experimental group (IVUS) steering group or control group (imaging) steering group.) Plan 10 centers in 200 men and women aged 18 and older patients, according to the American heart association and the United States The college of cardiology interventional treatment guidelines for the participants.

Each center recruiting number does not exceed 40% of the total plan recruitment.

ELIGIBILITY:
Inclusion Criteria:

-Clinical Inclusion (CI) Criteria: CI. Age > 18 years C2. Onset of STEMI > 30 minutes, but < 12 hours C3. ST segment elevation in at least 2 contiguous leads of≥ 1mm or newly developed LBBB on ECG C4. Willing and able to provide informed consent

* Angiographic Inclusion (AI) Criteria (visual estimate) AI1. Having at least one infarct-related coronary artery of which
* the Culprit lesion is suitable for stenting
* the reference diameter of culprit vessel is ≥ 2.5 mm but ≤ 4 mm
* the TIMI flow is ≤ 1 in culprit lesion segment prior to guide wire crossing AI2. No excessive tortuosity and calcification in the culprit lesion segment that allowing stent implantation

Exclusion Criteria:

* Clinical Exclusion (CE) Criteria CE1. Contraindicating to any concomitant study medications CE2. Having cardiogenic shock with hemodynamic instability CE3. A history of bleeding diathesis or known coagulopathy CE4. A history of cerebrovascular accident (CVA) or transient ischemic attack (TIA) within the past 6 months; or a history of intracranial tumor, aneurysm or arteriovenous malformations; or a history of active peptic ulcer or active gastrointestinal (GI) bleeding within the past 2 months; or planned major procedure within 6 weeks; or known platelet count < 100,000 /mm3 or Hb < 10 g/dL CE5. Planned surgery which may cause discontinuation of ADP-receptor antagonist CE6. Other serious illness (e.g., cancer) that may reduce life expectancy to less than 1 year CE7. Repeated MI within 7 days of hospitalization for acute MI
* Angiographic Exclusion (AE) Criteria (visual estimate) AE1. Bifurcated lesion unable to identify the culprit lesion AE2. The culprit lesion is located in the left main artery. AE3. Diffusive lesions without distinguishable culprit lesion AE4. Previous stent implantation in the culprit lesion segment or STEMI caused by stent thrombosis AE5. Likely CABG procedure within 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Jianan Wang, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- 2nd Affiliated Hospital, School of Medicine at Zhejiang University, Hangzhou, Zhejiang, China

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-04-15): https://cdn.clinicaltrials.gov/large-docs/58/NCT04929158/Prot_SAP_000.pdf
  • Informed Consent Form (2021-03-25): https://cdn.clinicaltrials.gov/large-docs/58/NCT04929158/ICF_001.pdf